CLINICAL TRIAL: NCT02384291
Title: Sinus Floor Elevation Using Alpha-Bio's GRAFT Natural Bovine Bone Versus Commercially Available Bone Graft. A Prospective Randomized Clinical Trial
Brief Title: Sinus Floor Elevation Using Alpha-Bio's GRAFT Natural Bovine Bone vs. Commercially Available Bone Graft
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Alpha - Bio Tec Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ABT-BG-01
Record Dates: First submitted 2015-02-26; First posted 2015-03-10 (Estimated); Last update posted 2019-07-16 (Actual); Status verified 2018-09

CONDITIONS: Sinus Floor Augmentation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Alpha-Bios GRAFT Natural Bovine Bone treatment (Experimental): Pure Hydroxyapatite ceramic mineral with high similarity to the human bone
  Interventions: Device: Alpha-Bio GRAFT Natural Bovine Bone
- natural bone substitute (Active Comparator): natural bone substitute material derived from the mineral portion of bovine bone
  Interventions: Device: natural bone substitute

INTERVENTIONS:
Device: Alpha-Bio GRAFT Natural Bovine Bone — Pure Hydroxyapatite ceramic mineral with high similarity to the human bone
  Arms: Alpha-Bios GRAFT Natural Bovine Bone treatment
Device: natural bone substitute — natural bone substitute material derived from the mineral portion of bovine bone
  Arms: natural bone substitute

SUMMARY:
This clinical study is designed to compare the regenerative outcome of using separately two different Xenografts during sinus floor augmentation.

Aim of this prospective randomized-controlled clinical trial is to compare the regenerative results of Alpha-Bio's GRAFT Natural Bovine Bone versus commercially available bone graft after two-step sinus floor elevations by clinical and histological analysis.

Clinical Parameters are wound healing parameters, radiological volume stability and implant survival rates. Histological parameters are based on a histomorphometrical analysis of trephine cores harvested in progress of implant bed preparation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who will present with a moderately or severely atrophic posterior maxilla with 1-6 mm residual alveolar bone will be selected for the study.
2. Men and women over the age of 18 years.
3. Patient has signed the Informed Consent.

Exclusion Criteria:

1. Chronic steroid therapy,
2. Uncontrolled diabetes,
3. Cardiovascular disease,
4. Past irradiation of head and neck
5. Maxillary sinus cysts,
6. Active chronic sinusitis,
7. Smoking more than ten cigarettes per day during the 3 months preceding this study .
8. Malignant disease in the 5 years preceding this study
9. Uncontrolled bleeding disorders such as: hemophilia, thrombocytopenia, granulocytopenia
10. Disease that compromise the immune system
11. Psychiatric disorder
12. Hypersensitivity to titanium, collagen or bovine bone.
13. Women who are pregnant or nursing.
14. Patients with non-treated periodontal disease.
15. Medical and/or general contraindications for intraoral surgical procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2014-05; Primary Completion 2019-12 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Histological bone formation following sinus floor augmentation [ evaluated by biopsies harvested from the implant sites] | 6 months

SECONDARY OUTCOMES:
Bone volume-stable results six months following augmentation procedures [ demonstrated by X-ray evaluation]. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Rothamel, Priv-Doz Dr., Principal Investigator — Department of Craniomaxillofacial and Plastic Surgery University Hospital of Cologne

REFERENCES:
- See also: Sponsor site — http://www.alpha-bio.net/global